CLINICAL TRIAL: NCT07155434
Title: Evaluation of Limited Trans Thoracic Echocardiography (L-TTE) by Non-Sonographers Using the UltraSight AI Guidance Software in Hypertrophic Obstructive Cardiomyopathy (HOCM) Patients Eligible for Mavacamten (Camzyos™) Treatment
Brief Title: ENABLE-HCM - AI-ENabled Echocardiography With Ultrasound Beyond the Echo Lab for Better HCM Imaging and Expanded Access
Status: Recruiting | Type: Observational
Sponsor: UltraSight (Industry)
Responsible Party: Sponsor
Other Study IDs: ULTRA-HCM-100
Record Dates: First submitted 2025-08-01; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hypertrophic Cardiomyopathy (HCM); Cardiac Imaging; Echocardiography; Mavacamten; Obstructive Cardiomyopathy, Hypertrophic
Keywords: hypertrophic cardiomyopathy; ultrasound; echocardiography; sonographer; monitoring; Guidance; software; UltraSight; image quality; REMS
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertrophic obstructive cardiomyopathy (HOCM) Patients Undergoing two Echo Exams: Hypertrophic obstructive cardiomyopathy (HOCM) patients who are eligible for or currently receiving Camzyos™ (mavacamten) will undergo two limited transthoracic echocardiography (LTTE) exams on the same day: one performed by a trained sonographer, and the other by a non-sonographer healthcare provider using the UltraSight Guidance Software. The study will compare the image quality and diagnostic agreement between the two sets of scans to evaluate the software's ability to support non-experts in performing cardiac ultrasound.

SUMMARY:
This study evaluates whether healthcare providers without specialized ultrasound training can use UltraSight's machine learning based Guidance Software to perform limited transthoracic echocardiography in patients with hypertrophic obstructive cardiomyopathy (HOCM), who are receiving or eligible for mavacamten (Camzyos™). Participants will undergo two heart scans on the same day, one by a non-sonographer using the software and one by a trained sonographer. The study aims to determine if the software-guided images are comparable in quality, with the goal of expanding access to heart monitoring for HCM patients.

DETAILED DESCRIPTION:
This study is evaluating whether healthcare providers without specialized ultrasound training can use UltraSight's Guidance Software to perform heart ultrasound exams (limited transthoracic echocardiography) in patients with hypertrophic obstructive cardiomyopathy (HOCM) who are receiving or eligible for treatment with Camzyos™ (mavacamten). The study aims to determine if the software-guided images are comparable to those taken by the sonographers, in quality. Participants will receive two echocardiography scans on the same day (one by a non-sonographer using UltraSight's Guidance Software and one by a sonographer), and the image quality will be reviewed by expert cardiologists. The study aims to increase patients' access to cardiac monitoring, especially for this patient population, by enabling more healthcare professionals to perform these echocardiography exams safely and effectively.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 years or over at the time of screening.
2. Willing and able to give written informed consent.
3. New York Heart Association (NYHA) Class I to III
4. Eligible to receive or currently receiving CamzyosTM per product labelling.

Exclusion Criteria:

1. Emergency (non-elective) admission within 24 hours prior to participating in the study.
2. Unable to lie down as required in all the classic positions for standard TTE exam: supine on back/left decubitus.
3. Subjects who had technically difficult exam in the past, due to body habitus, upon investigator's discretion.
4. Subjects with body mass index (BMI) above 40 kg/m2.
5. Subjects experiencing a known or suspected acute cardiac event.
6. Subjects with severe chest wall deformities as per previous medical records and physical examination.
7. Subjects who have undergone pneumonectomy.
8. Subjects whose anatomy does not lend itself to yield diagnosable echocardiography clips (i.e., situs inversus with dextrocardia, single ventricle anatomy due to congenital heart defect, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertrophic obstructive cardiomyopathy (HOCM) patients eligible for mavacamten (Camzyos™) treatment
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Agreement in Left Ventricular Ejection Fraction (LVEF) | 1 day
  To demonstrate agreement in echocardiography data between limited transthoracic echocardiography (LTTE) exams performed by non-sonographer healthcare professionals (HCPs) using the UltraSight Software and exams performed by trained sonographers. LVEF will be assessed using Simpson's Method and categorized into predefined groups. The expert cardiologists evaluating the LVEF will be blinded to the exam performer's identity.

SECONDARY OUTCOMES:
Agreement in Quality level of Specific Echocardiographic Views Between Non-Sonographer HCPs and Sonographers, using ACEP echocardiography images' quality scale | 1 day
  To demonstrate agreement in the quality of specific echocardiographic views obtained by non-sonographer healthcare professionals (HCPs) using the UltraSight Software compared to those obtained by trained sonographers. Quality will be assessed by blinded expert cardiologists using the 5-point American College of Emergency Physicians [ACEP] scale), for each of the following views: Parasternal Long-Axis (PLAX), Apical 2-Chamber (Apical 2C), Apical 3-Chamber (Apical 3C), Apical 4-Chamber (Apical 4C), Apical 5-Chamber (Apical 5C).
Number of participants with adverse events (AEs) as assessed by CTCAE v4.0 | 1 day
  The number of AEs, SAEs, and device related AEs will be captured as well as the number of subjects who discontinue due to an AE.

OTHER OUTCOMES:
Agreement in Left Ventricular Outflow Tract (LVOT) Gradient Categories Between Non-Sonographer HCPs and Sonographers | 1 day
  To assess agreement in the classification of LVOT gradient (in mmHg) during rest and Valsalva maneuver between exams performed by non-sonographer healthcare professionals using the UltraSight Software.

CONTACTS AND LOCATIONS:
Overall Officials: Milind Desai, MD., Principal Investigator — Cleveland Clinic, Cardiovascular Medicine Department
Locations (1):
- Cleveland Clinic, Cardiovascular Medicine Department, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not yet been finalized. While the study data will be de-identified, additional considerations such as the proprietary nature of the investigational device, regulatory strategy, and potential for future publications or secondary analyses are still being evaluated. IPD sharing may be considered after study completion and internal review.